CLINICAL TRIAL: NCT03430544
Title: A Randomized, Single-blind, Placebo-controlled Phase II Study to Assess the Effects of Cariprazine on Brain and Behavior in Subjects With Cocaine Use Disorder
Brief Title: Cariprazine Effects on Brain and Behavior in Cocaine Use Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment in final grant year, halted on-site research due to COVID-19 during NCE year.
Sponsor: Anna Rose Childress, Ph.D. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Anna Rose Childress, Ph.D., Research Professor of Psychology in Psychiatry, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 828585
Record Dates: First submitted 2018-01-29; First posted 2018-02-13 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Cocaine Use Disorder
Keywords: cariprazine; fMRI; D3 receptor; cocaine use disorder; urine
MeSH Terms: interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- 1.5 mg/d cariprazine (Experimental)
  Interventions: Drug: Cariprazine Oral Capsule [Vraylar]
- 3.0 mg/d cariprazine (Experimental)
  Interventions: Drug: Cariprazine Oral Capsule [Vraylar]

INTERVENTIONS:
Drug: Cariprazine Oral Capsule [Vraylar] — Cariprazine Groups (1.5 or 3mg/d): Cariprazine (VRAYLAR) capsules will be administered orally, once per day. Subjects in the 1.5mg group will receive 1 VRAYLAR capsule containing 1.5 mg cariprazine each day that study drug is administered. Subjects in the 3 mg group will be gradually titrated up to full dose: they will receive 1 VRAYLAR capsule containing 1.5mg cariprazine on the first and second days that study drug is administered and will receive 1 VRAYLAR capsule containing 3mg cariprazine each day for the rest of the medication period. The study medication period begins during the inpatient/induction phase and ends on the last day of outpatient treatment week 8 (approx. 10 weeks total). All VRAYLAR capsules will be over-encapsulated by the University of Pennsylvania Investigational Drug Services (IDS).
  Arms: 1.5 mg/d cariprazine; 3.0 mg/d cariprazine
Drug: Placebo oral capsule — PLACEBO Group: Visually identical placebo capsules will be supplied by the University of Pennsylvania Investigational Drug Service, with a dosing regimen matching the cariprazine groups.
  Arms: Placebo

SUMMARY:
This is a phase II, randomized, single-blind, placebo-controlled study to examine whether cariprazine (1.5 or 3 mg/d) 1) alters brain and/or behavioral responses to probes of reward and inhibition and 2) decreases cocaine use in individuals with cocaine use disorder. Subjects will be tested as inpatients during fMRI sessions. After the 2-week inpatient/medication induction phase, study medication will continue for 8 outpatient weeks, during which time cocaine use will be tracked. Subjects will be monitored during a 4-wk followup phase thereafter.

ELIGIBILITY:
Inclusion Criteria (limited):

1. An informed consent voluntarily signed and dated by the subject.
2. Physically healthy males and females with cocaine use disorder.
3. Ability to read at or above eighth grade level and speak, understand, and write in English.
4. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
5. Available for an inpatient stay, when applicable.

Exclusion Criteria (limited):

1. Certain psychological disorders that could put subjects at risk during participation in the study.
2. Certain lifetime or current medical disorders or conditions that could put subjects at risk during participation in the study.
3. Medical contraindications for MRI, when applicable.
4. Has received medication that could interact adversely with cariprazine within the time of administration of study agent based on the study physician's guidance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Primary fMRI outcome measure - BOLD signal change during visual cocaine vs. neutral cues. | Collected during fMRI scan 1, which takes place approximately 12-13 days after subject enrollment.
  The primary fMRI outcome is the extracted BOLD signal change during visual stimuli reminiscent of cocaine (i.e., cocaine cues) in an a priori circuit-level ROI.
Primary clinical outcome measure - percentage of urines cocaine-positive or missing during outpatient phase. | Urines are collected 3x per week during the 8 week outpatient phase.
  The primary clinical outcome is percentage of urines cocaine-positive or missing (assessed by urines positive for benzoylecgonine (BE), a metabolite of cocaine) throughout the outpatient treatment phase [Urines are counted as BE-positive if BE exceeds 300 ng/ml or if they are missing (no sample provided for a time point)].

SECONDARY OUTCOMES:
Secondary fMRI outcome measure - BOLD signal change during attempted inhibition of cue-triggered drug craving. | Collected during fMRI scan 2, which takes place approximately 13-14 days after subject enrollment.
  The secondary fMRI outcome is the extracted BOLD signal change during attempted inhibition of cue-triggered drug craving in an a priori ROI .
Attentional bias scores | Completed on approximately day 14-15 after subject enrollment.
  Attentional bias scores derived from reaction time (msec) during attentional bias task
Affective bias scores | Completed on approximately day 14-15 after subject enrollment.
  Affective bias scores derived from reaction time (msec) during affective bias task
Balloon Analogue Risk Task scores | Completed on approximately day 14-15 after subject enrollment.
  # of average adjusted pumps on BART
Go-NoGo Task scores | Completed on approximately day 14-15 after subject enrollment.
  # of errors of commission

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rose Childress, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States